

# **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Compassionate Access of the Miltenyi Device for CD34+ Cell Selection 2015-0295

| Study Chair: Elizabeth Shp | all |
|---|---|
| Participant's Name | Medical Record Number |
| | I authorization form for a research study. It includes a bre detailed description of procedures and risks is |

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

### STUDY SUMMARY

provided after the summary.

If you are reading and signing this form on behalf of a potential participant, please note: Any time the words "you," "your," "I," or "me" appear, it is meant to apply to the potential participant.

The goal of this expanded access study is to provide access to the Miltenyi device (which is used for CD34+ cell infusions) to patients who experience poor graft function after stem cell transplantation (SCT).

Your doctor believes that this is the best course of treatment for your present condition. Your doctor based this decision on a review of your medical history and consideration of available treatments.

**This is an investigational study.** The CD34 positive stem cell infusion to help boost cell counts is not FDA approved.

The CD34 positive cells may engraft (grow and multiply in your body), which may help your immune system and blood counts. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects,

potential expenses, and time commitment. If you take part in this study, you may experience increased infections. There may be other standard options.

You can read a list of potential side effects below in the Possible Risks section of this consent.

You may receive up to 2 CD34 positive stem cell infusions.

You and/or your insurance provider will be responsible for the costs of treatment.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive other therapy, if available. The study doctor will discuss the possible risks and benefits of these treatments. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

#### 1. STUDY DETAILS

Below is a detailed explanation of the therapeutic procedures that will be performed.

#### CD34 positive stem cells infusion

The CD34 positive stem cells are collected from a donor's blood. The blood cells go through CD34 (stem cell) selection process that collects the stem cells that are needed for the infusion. This process collects the early immune cells your body will need to regrow your immune system and makes sure that other cells will not be infused. This process will decrease (but not eliminate completely) the other types of cells. If you agree to receive this treatment, the CD34 cells will then be infused into your body.

The CD34 positive cells will be given by vein in either an inpatient or outpatient treatment area. The infusion will last about 10-30 minutes.

Before the infusion, you will receive Tylenol (acetaminophen) by mouth and Benadryl (diphenhydramine hydrochloride) by mouth or vein about 30-60 minutes before the infusion, depending on what the research team thinks is best. These drugs will be used to help lower the risk of side effects. If side effects occur during the infusion, the doses of the drugs may be adjusted (up or down) until the symptoms are gone. Also, if you have side effects during the infusion, you will be observed for 2 hours after it is given or until the symptoms have stopped completely (whichever is later). During this time, your blood pressure, heart rate, breathing rate, temperature, and the level of oxygen in your blood will be checked every 15-30 minutes.

About 4-6 weeks after the first infusion, you may receive an additional infusion, if your doctor thinks it is needed.

# **Clinic Visits**

One (1) time a week after the infusion, until your doctor thinks it is no longer clinically needed, you will have the following tests:

• Blood (about 1 teaspoon) will be drawn for routine tests.

• You will be checked for signs of graft versus host disease (GVHD). Symptoms of GVHD include skin rash, nausea, vomiting, diarrhea, and abnormal liver function.

Up to 200 patients will be enrolled on this treatment.

#### 2. POSSIBLE RISKS

While receiving treatment, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects that the treatment is known to cause. You should discuss these with the treating doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization or death.

#### CD34 Risks

The additional laboratory processing of stem cells may increase the risk of infection from the transplant. Because the antibody to CD34 is produced by mouse cells, it is possible that a person previously exposed to mouse proteins could have an allergic reaction to the stem cells. A small protein is used to remove antibodies from the cells, but this protein has not been associated with any known side effects. It is possible that an allergic reaction to this protein could occur. You will be monitored closely for any reaction to the stem cell infusion.

The CD34 stem cell infusion may cause allergic reactions and/or shortness of breath. The donor cells may fail to grow and multiply in your body (graft failure). If this occurs, you may have a high risk of infections and/or bleeding. You may need frequent blood transfusions. Graft failure can be treated with growth factors or a second transplant, but these treatments do not work all the time.

Once inside your body, the CD34 cells may react against your normal tissues, causing a reaction called GVHD. Acute GVHD may occur within the first several months after the transplant and may cause skin rash, diarrhea, and/or liver damage. Chronic GVHD may develop after the third month post-transplant and is considered a long-term complication involving the lungs, eyes, mouth, liver, skin, joints, digestive tract, and/or muscles.

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

This study may involve unpredictable risks to the participants.

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

# **Additional Information**

- 4. You may ask the study chair (Dr. Elizabeth Shpall, at 713-745-2161) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.
- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.

- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.

# **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and/or shared with other researchers and/or institutions for use in future research.

# Samples

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

#### Genetic Research

Research samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a

disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you. The same level of data protection that covers your individual data does not apply to summary results (when data from the whole study is combined).

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

# <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Miltenyi Biotec, Inc., The Center for International Blood and Marrow Transplantation Research (CIBMTR) and The National Marrow Donor Program (NMDP)
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

Any personal information that could identify you will be removed or changed before data are shared with other researchers or results are made public.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# CONSENT/AUTHORIZATION (Adult Participants Only)

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document.

| SIGNATURE OF PARTICIPANT | DATE |
|---|---|
| PRINTED NAME OF PARTICIPANT | |
| LEGALLY AUTHORIZED REPRESENTATIVE (LAR) | |
| The following signature line should only be filled out when the partithe capacity to legally consent to take part in the study and/or sinks or her own behalf. | • |
| SIGNATURE OF LAR | DATE |
| PRINTED NAME and RELATIONSHIP TO PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be perform protocol. | med under this |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIL A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. | DATE<br>R) |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his representative, using language that is understandable and appropriate I have fully informed this participant of the nature of this study benefits and risks and that the participant understood this explanation | oriate. I believe<br>y and its possible |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |

# PARENT/GUARDIAN PERMISSION I have read and understand the description of this research. I have had a chance to discuss the study and ask questions. My questions have been answered. I give permission for my child or ward to take part in this study. SIGNATURE OF PARENT/GUARDIAN DATE PRINTED NAME OF PARENT/GUARDIAN SIGNATURE OF PARENT/GUARDIAN DATE Signature of Other Parent (Optional, unless required by the IRB.) PRINTED NAME OF PARENT/GUARDIAN The IRB has determined that the signature of both parents is required. If not obtaining both parental signatures, please indicate reason below: Other parent is deceased, unknown, incompetent, or not reasonably available. Parent/Guardian signing above has sole legal responsibility for the care and custody of the child. **X** The IRB has determined that the signature of both parents is NOT required. WITNESS TO PARENTAL/GUARDIAN PERMISSION I was present during the explanation of the research to be performed under Protocol 2015-0295. The child participant was also present. In my opinion, the parent(s)/guardian provided permission for the child to participate in the research. SIGNATURE OF WITNESS TO THE PARENTAL/GUARDIAN DATE PERMISSION (OTHER THAN PARENT/GUARDIAN OR

PRINTED NAME OF WITNESS TO THE PARENTAL/GUARDIAN PERMISSION

MEMBER OF THE STUDY TEAM)

# **ASSENT OF MINOR**

(Entire section must be completed if the participant's intellectual age is at least 7 and less than 18 years. Participants with an intellectual age of 7 - 12 are not required to sign.)

| why not: |
|---|
| 1.) The participant's intellectual age is less than seven. |
| 2.) The participant dissented, but the participant's parent(s)/guardian felt that the intervention(s) or procedure(s) involved in the research hold out the possibility of a direct benefit that is important to the health and/or well being of the participant and is available only in the context of this research study3.) Other: |
| I have been told what I will be asked to do in this study. |
| I have been told that I do not have to be in this study. If I decide not to be in this study, no one will be mad at me. I may quit at any time, but if I do, I may need to take a different treatment. |
| I have had a chance to talk about the study and ask the study doctor questions. All of my questions have been answered. I agree to be in this study and do what I am asked to do so long as I want to stay in this study. I agree that the study doctor can put me on this study. By signing this paper, I am not giving up any of my legal rights. I have been given a copy of this document. |
| SIGNATURE OF MINOR (Age 13-17) DATE |
| PRINTED NAME OF MINOR |
| TRANSLATOR |
| I have translated the above informed consent as written (without additions or subtractions) intoand assisted the people (Name of Language) obtaining and providing consent by translating all questions and responses during the |
| consent process for this participant. |
| NAME OF TRANSLATOR SIGNATURE OF TRANSLATOR DATE |
| ☐ Please check here if the translator was a member of the research team. (If |

checked, a witness, other than the translator, must sign the witness line below.)